CLINICAL TRIAL: NCT01188382
Title: Reference Values of Cerebrospinal Fluid Outflow Resistance and Intracranial Pressure in Healthy Elderly
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Jan Malm, Dep Clinical Neuroscience
Other Study IDs: Hydrocephalus100
Record Dates: First submitted 2010-08-17; First posted 2010-08-25 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-06

CONDITIONS: Healthy Elderly
Keywords: Intracranial pressure; resistance; CSF outflow; elderly; reference value

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy elderly: Healthy elderly 60-82 years; Normal MRI; No psychiatric or neurological disorder and without signs of advanced atherosclerotic disease
  Interventions: Procedure: CSF dynamic investigation

INTERVENTIONS:
Procedure: CSF dynamic investigation

SUMMARY:
Objective. The intracranial pressure and cerebrospinal outflow resistance are essential parameters to describe the cerebrospinal fluid dynamic system. Outflow resistance effects intracranial pressure, pulse amplitudes, cerebrospinal fluid absorption as well as the compliance of the system. The objective of this study was to determine the reference values in the elderly.

Methods. Elderly people (60-82 years), considering themselves healthy, were recruited through an ad in the local paper. All were evaluated with a 3 Tesla magnetic resonance imaging apparatus. Subjects were eligible if they did not have any psychiatric or neurological disorder or signs of advanced atherosclerotic disease. Intracranial pressure and outflow resistance were determined by a constant pressure infusion method with the patient in the supine position. The study population consisted of 40 subjects (mean age 70 years; 23 women).

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 60-82 years

Exclusion Criteria:

* Psychiatric or neurological disorder or advanced atherosclerotic disease

Ages: 60 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy elderly
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
CSF outflow resistance

SECONDARY OUTCOMES:
Intracranial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Jan I Malm, PhD, MD, Principal Investigator — Umeå University
Locations (1):
- Dep Clincial Neuroscience, Umeå university, Umeå, Sweden

REFERENCES:
- [Derived] Jacobsson J, Qvarlander S, Eklund A, Malm J. Comparison of the CSF dynamics between patients with idiopathic normal pressure hydrocephalus and healthy volunteers. J Neurosurg. 2018 Nov 16;131(4):1018-1023. doi: 10.3171/2018.5.JNS173170. Print 2019 Oct 1. PMID 30497143
- See also: Web site of the Umeå hydrocephalus research group — http://www.hydrocephalus.se